CLINICAL TRIAL: NCT05478746
Title: Effects of Flourish HEC Vaginal Care System on Reduction of Pain in Women With Localized Provoked Vulvodynia
Brief Title: Effects of Flourish HEC on Localized Provoked Vulvodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaginal Biome Science (Other)
Collaborators: Evvy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPV0522
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Vulvodynia; Vestibulodynia; Vulvar Diseases; Vulvar Vestibulitis; Vulvar Pain
Keywords: Localized provoked vulvodynia; Vaginal microbiome; Probiotic; Lactobacillus
MeSH Terms: conditions — Vulvodynia; Vulvar Diseases; Vulvar Vestibulitis

STUDY DESIGN:
Intervention Model Description: Longitudinal open-label randomized controlled trial. Patients enrolled for 3 months in one of two concurrently enrolling groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine Care (Other): Participants enrolled in the control arm will undergo routine care for localized provoked vulvodynia according to the doctor's usual recommendations. These may include lidocaine cream, physical therapy, a compounded cream containing a blend of lidocaine, baclofen, amitryptyline, estradiol, testosterone, and bupivacaine, radiofrequency treatment, Naropin or botulinum toxin injections.
  Interventions: Other: Control - no intervention
- Flourish HEC (Experimental): Participants in the Flourish HEC arm will undergo routine care as described for the control arm. Instead of lidocaine cream, they will be given a 4% lidocaine gel (called "Relief", to be used up to 4x/day as needed) in an iso-osmotic, pH-balanced gel base. In addition, they will be given 3 products to use as described here, comprising the "Flourish HEC" kit (HEC = hydroxyethylcellulose, the principal gelling compound in the vaginal gel, to distinguish from the original Flourish kit using aloe).
  1. "Balance" - external vulvar wash to be used daily in the shower.
  2. "BioNourish" - vaginal moisturizing gel to be used every day before bed. Iso-osmotic and pH-adjusted with lactic acid to match healthy vaginal fluid.
  3. "BiopHresh" - vaginal homeopathic suppository with 7 vaginal probiotic strains, including Lactobacillus crispatus, to be used every 3rd day before bed.
  Interventions: Device: BioNourish, a component of the Flourish HEC kit

INTERVENTIONS:
Device: BioNourish, a component of the Flourish HEC kit — BioNourish is a vaginal moisturizing gel which obtained FDA 510k clearance in 2020. It is one component of the full system being tested. The main intervention is to use this kit to improve the vaginal microbiome.
  Arms: Flourish HEC
Other: Control - no intervention — No intervention; participants only receive routine care.
  Arms: Routine Care

SUMMARY:
This study is designed to determine whether improving the vaginal microbiome in women with localized provoked vulvodynia (LPV) may help improve pain better than routine care alone. The study randomizes women with LPV to either routine care or routine care plus a vaginal hygiene system designed to improve the vaginal microbiome. Women will be assessed for vaginal microbiome, vaginal pH, and pain before enrollment and after 6 weeks, and after 3 months. Women will also have pain assessed 2 weeks after enrollment without assessing vaginal microbiome and pH.

DETAILED DESCRIPTION:
Vulvodynia is a chronic pain condition affecting the tissues of the external genitalia in women. Localized provoked vulvodynia (LPV) is a specific subset of vulvodynia in which pain occurs upon touching specific sites on the vestibule (or, less commonly, another defined area), and which has been present for more than three months without a known cause. LPV is characterized both by allodynia (pain in response to a normally non-painful stimulus) and hyperalgesia (excessive pain response), leading to pain with sex, tampon use, and even with activities of daily life, such as sitting or wearing tight clothing.

It is becoming accepted that LPV occurs as a type of hypersensitivity to Candida and other antigens which occurs in susceptible women. LPV is an inflammatory condition with increased levels of B-cells, T-cells, and macrophages in tender areas vs. non-tender areas. The inflammatory process sparks neuroproliferation - growth of new nerve endings - which increases the density of nerve fibers in tender spots, especially in areas of lymphoid aggregates.

The vulvar and vaginal microbiomes are connected to each other; species found in one are often found in the other. In fact, Jayaram et al. showed that all vaginal species were also found on the vestibule, and the dominant vaginal species is also the dominant vestibular species, suggesting that vaginal secretions are a major contributor to the vestibular/vulvar microbiome. Three recent studies have examined the link between vulvodynia and the vaginal microbiome. Results vary by study, with one showing differences in the present vaginal microbiomes between women with vulvodynia and healthy women, and others not showing differences. These may be explainable by inclusion/exclusion criteria (two studies excluded women with active yeast infection; one study specified studying generalized, not localized, vulvodynia; while the others did not specify). But it is agreed that past alterations in the microbiome primed women for excessive pain in response to gentle stimuli.

Vaginal microbiome composition is known to affect immune activation in the vagina and vulva. Campisciano and colleagues showed that vaginal dysbiosis is associated with elevated levels of interleukin (IL)-1ra and IL-2, and lower levels of fibroblast growth factor (FGF)-beta and granulocyte-macrophage colony stimulating factor (GM-CSF) than observed in healthy vaginas. Another study by the same group reported associations between vaginal microbiome composition and IL-1alpha and IL-18. Doerflinger showed activation of the innate immune response by Lactobacillus iners (intermediate flora) and Fannyhessea vaginae (associated with bacterial vaginosis), but not L. crispatus (healthy flora). Of greatest relevance, Falsetta and colleagues investigated expression and activation of the toll-like receptor family and found seven of them to be expressed at higher levels in tissue biospies from tender spots in LPV than in control tissue, and that exposure to HIV increased expression of TLR7 expression and the downstream inflammatory molecule IL-6. Notably, no studies have examined whether improving the vaginal microbiome might lead to reductions in immune signaling in vulvodynia.

Taken together, it is reasonable to hypothesize that the constitution of the vaginal microbiome may influence the hypersensitivity to allergens that comprises the cause of LPV. It is also possible that improving the vaginal microbiome may reduce immune cell recruitment and activation, reducing pain. It is predicted that using sequencing-based technology, differences between the vaginal microbiomes of women with LPV and those without will be detectable. Furthermore, its is predicted that using an over-the-counter feminine hygiene system designed to support a healthy vulvovaginal microbiome will reduce pain in women with LPV over and above any reductions observed with standard-of-care treatment.

The investigators recently conducted an 11-week pilot study of similar design. Women with recurrent bacterial vaginosis (BV) were recruited to use the Flourish Vaginal Care System® for 11 weeks. Primary outcomes were vaginal fluid pH and whether or not women had BV recurrence. By the end of the study, the average vaginal fluid pH had fallen from mean (SD) of 4.54 (0.53) at week 0 to 4.08 (0.40) at week 11. At baseline, 30% of women had active BV. (These women were treated with standard of care oral metronidazole). The number of BV-positive women steadily declined until 5 weeks, at which point no woman had BV. There was no recurrence of BV in any woman through the end of the study. Women reported fewer vulvovaginal symptoms throughout the study. An ad hoc follow-up phone survey a year later showed that only one participant had a recurrence of BV since the end of the study. This study shows that the system we propose to use in the present study is able to effect positive changes in the vaginal microbiome.

A follow-up trial at the same center examining the vaginal microbiome using the same system for 6 months has shown very low recurrence rates, based on preliminary analysis, less than 20% in 6 months, compared with other studies showing 3-month recurrence rates of 43% or 62%. This study, which has completed data collection but has not yet been published, also showed that the vaginal microbiome was in a healthy or intermediate community state type (CST; not BV) during use of the system, though it took over 5 weeks of usage for one woman to move from a BV-like CST to a healthy CST. A similar study is underway using the "Flourish HEC" system - a nearly identical kit with a different vaginal moisturizing gel, gentler for those with sensitivities. To date, five participants are enrolled, and only the initial microbiome tests are available. However, study subjects are reporting that they are feeling good while using the system. It is this Flourish HEC system that will be tested in the present study. We emphasize that the vaginal care system is not intended to modify the body; it has no active drug components. Instead, it is a hygiene system that mimics the proper vaginal environment for a healthy microbiome to develop and thrive.

The investigators hypothesize that regular use of the Flourish HEC Vaginal Care System by women with LPV for three months will colonize the vagina and vulva with healthy bacteria, and that this will reduce inflammation, immune system activation, and neuroproliferation, ultimately reducing pain.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal cis women between ages 18 and 52 diagnosed with LPV via cotton swab test who have experienced symptoms for at least three months, and who do not have another diagnosis which may explain the pain.

Exclusion Criteria:

1. Known allergies or sensitivities to aloe or any other ingredients of the Flourish HEC Vaginal Care System
2. Individuals whose pain completely prevents application of intravaginal products (applicators similar in size to a tampon)
3. Individuals who are immunosuppressed or otherwise immunocompromised
4. Known allergy or sensitivity to metronidazole or fluconazole
5. Known active vaginal infection at the beginning of the study
6. Anyone who may have mental health disorders or trauma history triggered by answering questions related to vulvar or vaginal health, by pelvic exams, or self-application of vaginal products
7. Vulnerable populations: adults unable to consent, individuals who are not yet adults, pregnant or lactating women (or those attempting to become pregnant), and prisoners

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Vaginal microbiome in women with localized provoked vulvodynia (LPV) | Baseline
  Using whole-genome sequencing, all microbes present in the vaginal microbiome will be identified and reported for relative abundance.
Changes in the vaginal microbiome in women with localized provoked vulvodynia (LPV) with and without Flourish HEC | Baseline to 6 weeks.
  Using whole-genome sequencing, all microbes present in the vaginal microbiome will be identified and reported for relative abundance. Changes in these values from baseline to 6 weeks will be compared in women using or not using the Flourish HEC system.
Changes in the vaginal microbiome in women with localized provoked vulvodynia (LPV) with and without Flourish HEC | Baseline to 3 months.
  Using whole-genome sequencing, all microbes present in the vaginal microbiome will be identified and reported for relative abundance. Changes in these values from baseline to 3 months will be compared in women using or not using the Flourish HEC system.
Changes in the vaginal microbiome in women with localized provoked vulvodynia (LPV) with and without Flourish HEC | 6 weeks to 3 months.
  Using whole-genome sequencing, all microbes present in the vaginal microbiome will be identified and reported for relative abundance. Changes in these values from 6 weeks to 3 months will be compared in women using or not using the Flourish HEC system.
Pain intensity by cotton swab test | Baseline to 2 weeks to 6 weeks to 3 months.
  The PI will gently palpate the study participant at selected vulvar and extra-vulvar sites using a cotton swab; the participant will report pain on a scale of 0 (no pain) to 10 (most intense pain imaginable). Changes in pain intensity per location from baseline to 2 weeks, 6 weeks, and 3 months will be compared between women using and not using the Flourish HEC system.
Vulvovaginal symptoms questionnaire (VSQ) and addendum | Baseline to 2 weeks to 6 weeks to 3 months.
  Study participants responses to questions on the previously-validated VSQ and not-yet-validated additional questions will be collected on a 4-point Likert scale (0=not at all, 3 = all the time), except when questions are binary by nature. Change in question scores between timepoints will be compared between women who use and women who do not use the Flourish HEC system.

SECONDARY OUTCOMES:
Treatment escalation | Baseline to 2 weeks to 6 weeks to 3 months.
  A typical vulvodynia patient is started on a mild treatment, then escalated over time if symptoms do not improve. Treatment escalation will be compared between women who use and women who do not use the Flourish HEC system.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ojo-Carons, MD, Principal Investigator — EvoScient Gynecology
Locations (1):
- EvoScient Gynecology, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee Opinion No 673: Persistent Vulvar Pain. Obstet Gynecol. 2016 Sep;128(3):e78-e84. doi: 10.1097/AOG.0000000000001645. PMID 27548558
- [Background] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD), the International Society for the Study of Women's Sexual Health (ISSWSH), and the International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. Obstet Gynecol. 2016 Apr;127(4):745-751. doi: 10.1097/AOG.0000000000001359. PMID 27008217
- [Background] Paavonen J, Eschenbach DA. Localized Provoked Vulvodynia-An Ignored Vulvar Pain Syndrome. Front Cell Infect Microbiol. 2021 Jun 17;11:678961. doi: 10.3389/fcimb.2021.678961. eCollection 2021. PMID 34222047
- [Background] Liao Z, Chakrabarty A, Mu Y, Bhattacherjee A, Goestch M, Leclair CM, Smith PG. A Local Inflammatory Renin-Angiotensin System Drives Sensory Axon Sprouting in Provoked Vestibulodynia. J Pain. 2017 May;18(5):511-525. doi: 10.1016/j.jpain.2016.12.008. Epub 2017 Jan 3. PMID 28062309
- [Background] Tommola P, Unkila-Kallio L, Paetau A, Meri S, Kalso E, Paavonen J. Immune activation enhances epithelial nerve growth in provoked vestibulodynia. Am J Obstet Gynecol. 2016 Dec;215(6):768.e1-768.e8. doi: 10.1016/j.ajog.2016.07.037. Epub 2016 Jul 25. PMID 27457118
- [Background] Pagan L, Ederveen RAM, Huisman BW, Schoones JW, Zwittink RD, Schuren FHJ, Rissmann R, Piek JMJ, van Poelgeest MIE. The Human Vulvar Microbiome: A Systematic Review. Microorganisms. 2021 Dec 12;9(12):2568. doi: 10.3390/microorganisms9122568. PMID 34946169
- [Background] Jayaram A, Witkin SS, Zhou X, Brown CJ, Rey GE, Linhares IM, Ledger WJ, Forney LJ. The bacterial microbiome in paired vaginal and vestibular samples from women with vulvar vestibulitis syndrome. Pathog Dis. 2014 Dec;72(3):161-6. doi: 10.1111/2049-632X.12197. Epub 2014 Jul 10. PMID 24961922
- [Background] Park SY, Lee ES, Lee SR, Kim SH, Chae HD. Vaginal Microbiome Is Associated With Vulvodynia, Vulvar Pain Syndrome: A Case-Control Study. Sex Med. 2021 Apr;9(2):100314. doi: 10.1016/j.esxm.2020.100314. Epub 2021 Feb 27. PMID 33652201
- [Background] Mitchell CM, Watson L, Mitchell AJ, Hyrien O, Bergerat A, Valint DJ, Pascale A, Hoffman N, Srinivasan S, Fredricks DN. Vaginal Microbiota and Mucosal Immune Markers in Women With Vulvovaginal Discomfort. Sex Transm Dis. 2020 Apr;47(4):269-274. doi: 10.1097/OLQ.0000000000001143. PMID 32044865
- [Background] Bedford L, Parker SE, Davis E, Salzman E, Hillier SL, Foxman B, Harlow BL. Characteristics of the vaginal microbiome in women with and without clinically confirmed vulvodynia. Am J Obstet Gynecol. 2020 Sep;223(3):406.e1-406.e16. doi: 10.1016/j.ajog.2020.02.039. Epub 2020 Mar 2. PMID 32135142
- [Background] Campisciano G, Zanotta N, Licastro D, De Seta F, Comar M. In vivo microbiome and associated immune markers: New insights into the pathogenesis of vaginal dysbiosis. Sci Rep. 2018 Feb 2;8(1):2307. doi: 10.1038/s41598-018-20649-x. PMID 29396486
- [Background] De Seta F, Campisciano G, Zanotta N, Ricci G, Comar M. The Vaginal Community State Types Microbiome-Immune Network as Key Factor for Bacterial Vaginosis and Aerobic Vaginitis. Front Microbiol. 2019 Oct 30;10:2451. doi: 10.3389/fmicb.2019.02451. eCollection 2019. PMID 31736898
- [Background] Doerflinger SY, Throop AL, Herbst-Kralovetz MM. Bacteria in the vaginal microbiome alter the innate immune response and barrier properties of the human vaginal epithelia in a species-specific manner. J Infect Dis. 2014 Jun 15;209(12):1989-99. doi: 10.1093/infdis/jiu004. Epub 2014 Jan 7. PMID 24403560
- [Background] Falsetta ML, Foster DC, Woeller CF, Pollock SJ, Bonham AD, Piekna-Przybylska D, Maggirwar SB, Haidaris CG, Phipps RP. Toll-Like Receptor Signaling Contributes to Proinflammatory Mediator Production in Localized Provoked Vulvodynia. J Low Genit Tract Dis. 2018 Jan;22(1):52-57. doi: 10.1097/LGT.0000000000000364. PMID 29271858
- [Background] Chidawanyika T, Yi CHC, Kelly-Martin R, Cleland J, DuPriest E. Clinical trial to survey results of Flourish vaginal care system for recurrent BV [A80]. Obstet Gynecol. 2022;139:24S. doi:10.1097/01.AOG.0000826648.49549.01
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Sobel JD, Schmitt C, Meriwether C. Long-term follow-up of patients with bacterial vaginosis treated with oral metronidazole and topical clindamycin. J Infect Dis. 1993 Mar;167(3):783-4. doi: 10.1093/infdis/167.3.783. No abstract available. PMID 8440952